CLINICAL TRIAL: NCT02620748
Title: Use of Intravenous Tranexamic Acid During Myomectomy: A Randomized Double-Blind Placebo Controlled Trial
Brief Title: Use of Intravenous Tranexamic Acid During Myomectomy
Acronym: TA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 091454
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2019-01

CONDITIONS: Hemorrhage/Blood Loss During Myomectomies; Fibroids
MeSH Terms: conditions — Hemorrhage; Leiomyoma | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid (Experimental): This arm will receive an injection of Tranexamic Acid
  Interventions: Drug: Tranexamic Acid
- Saline (Placebo Comparator): This arm will receive an injection of Saline Solution
  Interventions: Other: Saline Solution

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic Acid
Other: Saline Solution
  Arms: Saline

SUMMARY:
The purpose of this study is to determine the effect of the early administration of intravenous (IV) Tranexamic acid (TA) on perioperative bleeding (as defined by measured intraoperative estimated blood loss (EBL), change in pre and post-operative hemoglobin (Hb), and frequency of blood transfusions) in women undergoing a myomectomy.

DETAILED DESCRIPTION:
Worldwide about 25% of women will develop uterine leiomyomas. Most myomas are asymptomatic however 20 to 25% of women with myomas develop symptoms, such as heavy menstrual bleeding, requiring treatment. For women failing medical management and desiring to preserve fertility and/or their uterus, surgical removal of fibroids (myomectomy) is the major option. Myomectomy is associated with both short and long-term complications, most significantly, hemorrhage and need for conversion to hysterectomy in 2% of cases, need for a blood transfusion in up to 20% of cases, prolonged postoperative stay, and can be potentially life-threatening. As such, various treatments have been suggested to decrease blood loss during myomectomy including pharmacologic manipulation of the coagulation cascade using agents such as tranexamic acid (TA). Despite the many described methods to reduce intraoperative bleeding, massive hemorrhage during myomectomy remains a significant challenge to gynecologic surgeons.

TA is a synthetic lysine derivative with antifibrinolytic activity that helps prevent clot break down. It is currently clinically used widely to stop heavy menstrual bleeding and many of the investigators' myomectomy patients are taking oral TA around the time of surgery. Systematic reviews of randomized control trials (RCTs) including over 25,000 patients of tranexamic acid in elective surgery showed that it reduced the risk of a blood transfusion by 34% (relative risk (RR) 0.61, 95% confidence interval (CI) 0.53 to 0.70) without an increased risk in venous thrombus embolus (VTE) or other adverse perioperative outcomes (Henry, 2011). Only one RCT has studied the use of TA during gynecologic surgery. This study was a randomized double blind placebo controlled trial of intravenous TA 10 mg/kg (maximum 1g) versus placebo during myomectomy procedures. Although there was a 63 ml decrease in postoperative blood loss (p<0.01), no significant difference was found between the two groups in terms of perioperative blood loss, change in hemoglobin, or rate of allogeneic blood transfusions. Further studies are needed with different dosing administration to confirm the true role of TA in the reduction of blood loss during myomectomy.

If a difference is seen, the results of future publications would directly impact clinical care locally and abroad, as few methods currently exist to prevent hemorrhage during myomectomy procedures.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing laparoscopic, robotic or abdominal myomectomy
* fibroid burden meeting the following criteria based on ultrasound imaging: Fibroids greater than or equal to 10 cm Intramural or Broad Ligament Fibroid greater than or equal to 6 cm Number of fibroids greater than or equal to 5 cm

Exclusion Criteria:

* Medical history of the following: thromboembolic disease, ischemic heart disease, malignancy, hematuria, liver disease, chronic kidney disease or subarachnoid hemorrhage
* pregnant women
* women who are nursing
* women with active thrombotic or thromboembolic disease
* women with history of intrinsic risk of thrombosis or thromboembolism
* hypersensitivity to Tranexamic Acid

Concurrent use of:

* combination of hormonal contraception
* factor IX complex concentrates
* Anti-inhibitor coagulant concentrates
* all-trans retinoic acid

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Blood Loss | At time of Surgery
  the volume of blood loss will be measured at end of surgery.

SECONDARY OUTCOMES:
change in pre-operative and immediately post-operative hemoglobin | At time of Surgery
frequency of blood transfusions | At time of Surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Faculty Associates, Washington D.C., District of Columbia, United States